CLINICAL TRIAL: NCT03549728
Title: Effect of Granulocyte Colony-stimulating Factor on Clinical Pregnancy Rate in Patients With Endometriosis Undergoing In-vitro Fertilization After Recurrent Implantation Failure
Brief Title: Effect of Granulocyte Colony-stimulating Factor on Clinical Pregnancy Rate in Patients With Endometriosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amira Magdi Guergues Selim (Other)
Responsible Party: Sponsor-Investigator, Amira Magdi Guergues Selim, Resident of obstetrics and gynecology, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2808
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Recurrent Implantation Failure; Endometriosis
Keywords: endometriosis; granulocyte colony-stimulating factor; recurrent implantation failure
MeSH Terms: conditions — Endometriosis | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the effect of granulocyte colony-stimulating factor on clinical pregnancy rate in patients with endometriosis undergoing in-vitro fertilization after recurrent implantation failure.
Who Masked: Participant, Care Provider, Investigator
Masking Description: : Eighty eight envelopes will be numbered serially and in each envelope the corresponding letter which denotes the allocated group will be put according to randomization table. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside into group A or B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A (N=44): women will receive intrauterine infusion of granulocyte colony-stimulating factor on the day of ovum-pick up during IVF cycle.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor
- Group B (Placebo Comparator): Group B (N=44): women will receive placebo intrauterine infusion of normal saline on the day of ovum-pick up during IVF cycle.
  Interventions: Procedure: Intrauterine infusion of normal saline

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor — In group A, at the day of oocyte retrieval, after oocytes collection, 30 mU (300 mcg/0.5 ml) of G-CSF (NeupogenTM, Filgastrim, Amgen Inc., Thousand Oaks, CA, USA) was administered by slow transcervical intrauterine infusion with IUI catheter (AINSEGREY, RIMOS, Italy). In controls, normal saline was used for intrauterine infusion instead of G-CSF.
  Other Names: Neupogen; Filgrastim
  Arms: Group A
Procedure: Intrauterine infusion of normal saline — In group B (controls), normal saline will be used for intrauterine infusion instead of granulocyte colony-stimulating factor on the day of oocyte retrieval.
  Arms: Group B

SUMMARY:
The aim of this study is to evaluate the effect of granulocyte colony-stimulating factor on clinical pregnancy rate in patients with endometriosis undergoing in-vitro fertilization after recurrent implantation failure.

DETAILED DESCRIPTION:
* Type of Study: A randomized double-blind controlled trial.
* Study Setting: IVF unit in Maternity Hospital of Ain Shams University.
* Study Population: A total of 88 women with endometriosis will be enrolled in the study divided into two groups:

  * Group A (N=44): women will receive intrauterine infusion of G-CSF on the day of ovum-pick up during IVF cycle.
  * Group B (N=44): women will receive placebo intrauterine infusion of saline on the day of ovum-pick up during IVF cycle.
* Allocation and Concealment: Eighty eight envelopes will be numbered serially and in each envelope the corresponding letter which denotes the allocated group will be put according to randomization table. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside
* Randomization Table:

SN Group SN Group SN Group SN Group SN Group SN Group SN Group SN Group

1. A 12 A 23 B 34 B 45 A 56 A 67 B 78 B
2. B 13 A 24 A 35 B 46 A 57 A 68 B 79 A
3. B 14 A 25 B 36 A 47 B 58 B 69 B 80 A
4. B 15 A 26 A 37 A 48 B 59 B 70 A 81 B
5. A 16 A 27 B 38 B 49 B 60 B 71 B 82 A
6. A 17 A 28 A 39 B 50 B 61 A 72 B 83 B
7. A 18 B 29 B 40 B 51 A 62 B 73 A 84 B
8. B 19 B 30 A 41 A 52 A 63 A 74 B 85 B
9. A 20 A 31 A 42 B 53 A 64 B 75 A 86 B
10. A 21 B 32 A 43 A 54 B 65 B 76 B 87 A
11. A 22 B 33 B 44 A 55 A 66 B 77 A 88 A

    * Sample Size: 88 patients, 44 in group A (the cases) and 44 in group B (the controls).
    * Sample Justification:

The required sample size was calculated using the G*Power Software (Universitӓt Düsseldorf, Germany).

The primary outcome measure is the clinical pregnancy rate. Currently, there is no adequate information regarding the effect of granulocyte colony-stimulating factor on clinical pregnancy rate in patients with endometriosis undergoing in-vitro fertilization; therefore, the present exploratory study would target an effect size that could be clinically relevant.

So, it is estimated that the inclusion of 44 patients in each of the 2 study groups (total, 88 patients) would achieve a power of 80% (type II error, 0.2) to detect a statistically significant difference between the 2 groups as regards the clinical pregnancy rate for a medium effect size corresponding to a w coefficient of 0.3 using a two-sided chi-squared test with 1 degree of freedom and the targeted test confidence set at a level of 95% (type I error. 0.05). The effect size (w) is calculated as follows:

w = , where is the chi-squared statistic and N is the total sample size (Chow et al., 2003).

The targeted effect size of w = 0.3 has been selected as it could be regarded as a clinically relevant difference to seek in this exploratory study.

* Ethical Considerations: A written informed consent will be obtained from all participants prior to screening and enrollment. Participants will participate voluntarily in the research and their confidentiality will be respected. Benefits from participation in the research will be explained to all participants. Participation in the research will cause no harm to participants after approval of research ethical committee.
* Study Procedures:

All participants will be subjected to the following:

A) Detailed medical history including:

* Personal history
* Menstrual history
* Past and obstetric history

B) Physical examination:

After history taking and fulfillment of both inclusion and exclusion criteria, clinical examination will be done including: general abdominal and pelvic examination.

C) Laboratory investigations:

Routine investigations including: fasting and postprandial blood sugar and complete blood count.

D) Induction of ovulation:

* On day 3 of spontaneous cycles, all patients will have basal hormonal profile (FSH, LH, E2, TSH and prolactin).
* Transvaginal (TV) ultrasound (U/S) on day 3 of non-stimulated cycles will be done by transvaginal probe of 5-9 MHZ. Any patient found to have uterine abnormalities will be excluded.
* Ovarian hyper stimulation protocol will be held according to a long GnRH agonist protocol starting from midluteal phase by daily subcutaneous injection of triptoreline acetate (Decapeptyl 0.05 mg, Ferring Pharmaceutical, Kid, Germany). Then on day 3 of next cycle ovarian hyper stimulation will be started by daily injection of HMG (Menogon 75 lU/amp "Ferring Pharmceutical, Kid, Germany "or Merional 75 IU/amp" IBSA, Switzerland"). The starting dose of gonadotropines will be prescribed according to the age and body weight of the subjects, then the dose will be adjusted according to the ovarian response that will be assessed by transvaginal folliculometry which will be done on cycle day six.
* According to the ovarian response, every other day TV U/S will be performed and at the moment when the leading follicle reaches 16mm, daily TV U/S will be performed till the largest follicle reach a diameter of >18mm. The maximum duration of HMG will not be allowed to exceed day 16.
* HCG (Choriomon 10,000 lU/amp. "IBSA, Switzerland") will be administered for triggering ovulation.

E) Sonography:

Transvaginal sonography will be performed in the day of HCG administration to measure endometrial thickness and pattern.

The endometrium pattern will be classified as:

* Proliferative when echogenicity is hypo echoic in relation to the myometrium.
* Peri-ovulatory when it is trilaminar.
* Secretory when it is hyperechoic.

F) Ovum pick up:

* 36 hours after HCG injection, the transducer will be connected to the ultrasound system. The direction of the guide beam will be checked. The puncturing needle will be connected to an aspiration apparatus attached by a fixation ring to the front and rear ends of the vaginal transducer, thereby defining the direction of puncture corresponding to the guide beam on the ultrasound image.
* The aspiration will be checked using test tubes. The uterus, both ovaries and iliac vessels will be identified by the visualization in both planes. The distance between the upper pole of the vagina and the ovary will be closely evaluated (care will be taken to avoid intestinal or vascular interposition).
* Depth localization of the closest accessible follicle (distance from the upper vaginal pole to the center of the follicle) will be done. Needle will be pushed forcefully to the center of the follicle (Aspiration pressure 90-100mmHg).

G) IVF- ICSI:

- Intracytoplasmic sperm injection will be performed on metaphase II oocytes using the direct penetration technique, fertilization results will be assessed 16 to 19 hours after ICSI. Fertilization will be considered normal by the presence of two pronuclei. Oocyte degeneration will be identified by collapse of cytoplasmic contents and separation from the zona. Failed fertilization will be defined by the absence of the pronuclei.

H) Embryo transfer:

* Embryo transfer will be done on day 5 using cook catheter under ultrasound guide at a distance about 1-1.5 cm from the fundus by the same gynecologist.
* Number of embryos transferred 2-3 embryos.

I) Finally:

A serum βhCG will be performed 12 days after embryo transfer and repeated after 48h. followed by US 6 weeks after embryo transfer.

* Study Interventions: In G-CSF group at the day of oocyte retrieval, after oocytes collection, 30 mU (300 mcg/0.5 ml) of G-CSF (NeupogenTM, Filgastrim, Amgen Inc., Thousand Oaks, CA, USA) was administered by slow transcervical intrauterine infusion with IUI catheter (AINSEGREY, RIMOS, Italy). In controls, normal saline was used for intrauterine infusion instead of G-CSF.
* Statistical Analysis: Data will be analyzed using IBM© SPSS© Statistics version 22 (IBM© Corp., Armonk, NY). Normally distributed numerical data will be presented as mean and SD, and skewed data as median and interquartile range. Qualitative data will be number and percentage. Comparison of normally distributed numerical data will be done using the unpaired t test. Skewed data will be compared using the Mann-whitney test. Categorical data will be compared using the Pearson chi-squared test or fisher's exact test, if appropriate. A two-sided p-value ˂0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Cases of infertility, older than 20 years of age and not older than 40 years.
* Body mass index (BMI): 20-29.
* Women diagnosed with endometriosis (diagnosis based on ultrasound or laparoscopy or both)
* Recurrent implantation failure (failure to conceive following two embryo transfer cycles, or cummulative transfer of >10 good quality embryos)
* Normal ovulatory cycles (as proven by folliculometry and/or mid luteal serum progesterone), good ovarian reserve (as proven by early follicular FSH and AMH)
* Normal uterine cavity as assessed by ultrasonography, hysterosalpingography, or hysteroscopy
* Normal hormonal profile (serum PRL, TSH, thyroid hormone)
* Normal semen analysis of the partner
* Infertility after one year of unprotected intercourse
* High-quality embryos were transplanted

Exclusion Criteria:

* Congenital or acquired uterine abnormalities (e.g. septate, bicornuate, fibroid uterus, uterine polyp & Asherman Syndrome)
* Congenital or acquired tubal abnormalities (e.g. hydrosalpinx or pyosalpinx)
* Contraindication for G-CSF (renal disease, sickle cell disease, or malignancy history, upper respiratory tract infection, pneumonia, or chronic neutropenia)
* Thrombophilia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Chromosomally 46XX
Enrollment: 88 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 5-6 weeks from the day of embryo transfer
  The primary outcome measure is the clinical pregnancy rate defined as the observation of gestational sac on transvaginal ultrasound examination three weeks after positive serum βhCG.

SECONDARY OUTCOMES:
Chemical pregnancy rate | 12 days after embryo transfer
  Positive serum βhCG test
Implantation rate | 6 weeks after embryo transfer
  The number of gestational sacs divided by the number of transferred embryos in each group
Ongoing pregnancy rate | 12 weeks of pregnancy
  The presence of fetal heart activity by ultrasonography after 12 weeks of pregnancy
Miscarriage rate | Before 20 weeks of pregnancy
  The number of miscarriages before 20 weeks gestation per number of women with positive βhCG test